CLINICAL TRIAL: NCT00450463
Title: A Randomized Phase II Trial Combining Vaccine Therapy With PROSTVAC/TRICOM and Flutamide vs. Flutamide Alone in Men With Androgen Insensitive, Non-Metastatic (D0.5) Prostate Cancer
Brief Title: Vaccine Therapy With PROSTVAC/TRICOM and Flutamide Versus Flutamide Alone to Treat Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ravi A. Madan, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 070107; 07-C-0107
Record Dates: First submitted 2007-03-20; First posted 2007-03-22 (Estimated); Results first posted 2018-11-26 (Actual); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Prostate Cancer
Keywords: Immunotherapy; Hormonal Therapy; Combination Therapy; Prostate Specific Antigen; Immunoassay; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — sargramostim; Granulocyte-Macrophage Colony-Stimulating Factor; Flutamide; PROSTVAC; Benchmarking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Flutamide Alone (Active Comparator): Patients receive flutamide orally 3 times a day on days 1-28. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity. After 3 months of treatment, patients who do not develop clinical progression, but develop biochemical recurrence (e.g., rising prostatic specific antigen (PSA) levels) without metastatic disease (as evidenced on scans), may receive vaccine treatment as defined in arm II beginning 4 weeks after flutamide therapy is discontinued.
  Interventions: Drug: Flutamide (Eulexin)
- Flutamide + Vaccine + Sargramostim (Experimental): Patients receive flutamide orally 3 times a day on days 1-28. Patients also receive recombinant vaccinia PSA vaccine subcutaneously (SC) on day 1 of course 1 only and recombinant fowlpox PSA vaccine SC on day 1 of all subsequent courses. Patients receive sargramostim (GM-CSF) SC on days 1-4. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity. After 3 months of treatment, patients who do not develop clinical progression, but develop biochemical recurrence (e.g., rising PSA levels), discontinue flutamide but may continue to receive vaccine treatment.
  Interventions: Drug: Sargramostim (GM-CSF, Leukine); Drug: Flutamide (Eulexin); Biological: PROSTVAC-F/ TRICOM; Biological: PROSTVAC-V/TRICOM

INTERVENTIONS:
Drug: Sargramostim (GM-CSF, Leukine) — A recombinant human granulocyte-macrophage colony stimulating factor (GM-CSF) produced by recombinant deoxyribonucleic acid (DNA) technology in yeast Saccharomyces cerevisiae). Sargramostim is a 127 amino acid glycoprotein, altered from the native, natural human GM-CSF molecule; the position 23 arginine has been replaced with a leucine to facilitate the expression of the protein in yeast.
  Other Names: GM-CSF
  Arms: Flutamide + Vaccine + Sargramostim
Drug: Flutamide (Eulexin) — Orally administered, nonsteroidal, competitive antagonist of testosterone and other androgens at androgenic receptors and may alter the nuclear translocation of the androgen/receptor complex.
  Other Names: Eulexin
Biological: PROSTVAC-F/ TRICOM — A recombinant fowlpox virus vector vaccine containing the genes for human PSA and three costimulatory molecules.
  Other Names: PROSTVAC-F (rilimogene galvacirepvec/rilimogene glafolivec)/TRICOM (triad of costimulatory molecules
  Arms: Flutamide + Vaccine + Sargramostim
Biological: PROSTVAC-V/TRICOM — A recombinant vaccinia virus vector vaccine containing the genes for human prostatic specific antigen (PSA) and three co-stimulatory molecules.
  Arms: Flutamide + Vaccine + Sargramostim

SUMMARY:
Background:

* Flutamide is an approved drug for prostate cancer that blocks the effects of testosterone on prostate cancer cells and may slow the progression of the disease.
* The vaccine in this study consists of a priming vaccine called PROSTVAC (rilimogene galvacirepvec/rilimogene glafolivec) -V/TRICOM (triad of costimulatory molecules), made from vaccinia virus, and a boosting vaccine called PROSTVAC-F/TRICOM, made from fowlpox virus. DNA (Deoxyribonuceic acid) is inserted into the priming and boosting vaccine viruses to cause production of proteins that enhance immune activity and also to produce prostate specific antigen (PSA) a protein that is normally produced by the patients tumor cells.
* GM-CSF (granulocyte macrophage colony stimulating factor), given along with the vaccine, is a chemical that boosts the immune system. It is used in this study to try to increase the usefulness of the vaccine by increasing the number of immune cells at the vaccination site.

Objectives:

-To determine if treatment with a prostate cancer vaccine plus flutamide is more effective than flutamide alone in delaying disease progression in patients with prostate cancer.

Eligibility:

* Patients 18 years of age and older with androgen-insensitive prostate cancer that has not spread beyond the prostate gland.
* Patients with a rising PSA (prostatic specific antigen) who have already been treated with anti-iandrogen therapy (either bicalutamide or nilutamide).

Design:

* There are two treatment groups in this study. Group A receives only flutamide; group B receive flutamide plus vaccine.
* Patients in both groups receive flutamide by mouth three times a day.
* Patients in group B receive PROSTVAC-V/TRICOM on day 1 and PROSTVAC-F/TRICOM on day 29 and again every 4 weeks. All vaccines are given as injections under the skin.
* Patients have blood tests for PSA levels every month and scans every 3 months until the disease worsens.
* After 3 months of therapy, patients receiving in group A (flutamide alone) may cross over to receive vaccine if they develop a rising PSA and scans show no sign of disease spread. Patients in group B (flutamide plus vaccine) stop flutamide and may continue vaccine therapy. At this point patients may continue to receive treatment until the disease progresses or PSA levels rise....

DETAILED DESCRIPTION:
Background:

* There is no standard of care for prostate cancer patients progressing on hormone therapy with a rising serum PSA (prostatic specific antigen) level without evidence of metastatic disease.
* We have completed a phase II trial in which men with this stage of disease were randomized to receive a pox vector PSA vaccine vs. the antiandrogen nilutamide.
* The median time to treatment failure on nilutamide was 7.6 months.
* 12 patients on the vaccine arm had nilutamide added at the time of PSA progression.
* The median time for treatment failure after the addition of nilutamide was 13.9 months, for a total of 25.9 months from initiation of vaccine therapy.
* This suggests that the combination of hormone therapy with vaccine therapy may lead to an improved clinical benefit compared to hormone therapy alone.
* Due to the increased toxicity of nilutamide compared to other antiandrogens and the patients prior exposure to bicalutamide therapy, we plan to use flutamide as a second line hormonal manipulation in the below study.

Objectives (Primary):

-To determine if use of a combination of vaccine plus flutamide may be associated with a trend toward improvement in time to treatment failure compared to flutamide alone.

Eligibility:

* Must have non metastatic androgen insensitive prostate cancer with a rising PSA with castrate levels of testosterone and no evidence of metastatic disease on CT (computed tomography) scan or bone scan.
* Hgb (hemoglobin) greater than or equal to 9 g/dL.
* Lymphocyte count greater than or equal to 500/mm(3).
* Hepatic function: Bilirubin less than or equal to 1.5 mg/dL, OR patients with Gilbert's syndrome, a total bilirubin less than or equal to 3.0 mg/dL, AST (aspartate aminotransferase) and ALT (alanine aminotransferase) less than 2.5 times upper limit of normal

Design:

-Flutamide will be administered at a dose of 250 mg PO (by mouth) tid (three times a day) every day in both arms A and B.

rV-PSATRICOM will be administered s.c. (subcutaneous) on day 1 in Arm B.

rF-PSATRICOM will be administered s.c. on day 29 & every 4 weeks in Arm B.

* For patients with declining PSA no restaging will be done unless they develop symptoms consistent with metastatic disease.
* For patients with rising PSA, once 2 consecutive PSA rises are seen, a CT will be done at their next scheduled visit. They will then be re-staged (CT and bone scans) at 3 month intervals as long as PSA continues to rise.
* After 3 months of therapy, patients receiving the flutamide alone (arm A) may cross over to receive vaccine if they develop a rising PSA and scans are without metastatic disease. The vaccine may commence 4 weeks after flutamide is stopped if the PSA continues to rise. If there is an antiandrogen withdrawal response (a decline in PSA 28 days after the discontinuation of flutamide), PSA serum levels will be checked every 28 days and vaccine may commence when the serum PSA levels begin to rise (if scans are negative for metastatsis). Patients on arm B will have flutamide discontinued and may continue vaccine therapy. At this point patients may continue to receive treatment on study until the development of disease on scans or a second occurrence of clinical progression.
* Patients who have been on study for 2 years or more with stable disease and who are not getting vaccine, clinic visits may be scheduled every 8 weeks. (Patients receiving monthly vaccine will continue to have monthly visits.)
* For patients who have stable disease and attend clinic every 8 weeks, once 2 consecutive PSA rises are seen, a CT and bone scan will be done at their next visit in 4 weeks. They will then be restaged (CT and bone scans) at 3 month intervals as long as PSA continues to rise.

ELIGIBILITY:
* INCLUSION CRITERIA:

A. Histopathological documentation of prostate cancer confirmed in the Laboratory of Pathology at the: National Institutes of Health (NIH) Clinical Center prior to starting this study. If no pathologic specimen is available, patients may enroll with a pathologists report showing a histologic diagnosis of prostate cancer and a clinical course consistent with the disease.

B. Must have non-metastatic androgen insensitive prostate cancer with a rising PSA (prostatic specific antigen) with castrate levels of testosterone and no evidence of metastatic disease on CT (computed tomography) scan or bone scan. A rising PSA is defined as two consecutively rising PSA levels, separated by at least 1 month apart, with the last measurement that is greater than 1ng/ml. Patients on nilutamide therapy must undergo nilutamide withdrawal for at least 4 weeks and still show evidence of a rising PSA. Following treatment with bicalutamide, patients must undergo withdrawal for at least 6 weeks and still show evidence of a rising PSA.

C. Life expectancy greater than or equal to 6 months.

D. ECOG (Eastern Cooperative Oncology Group) performance status of 0-1.

E. No systemic steroid or steroid eye drop use within 2 weeks prior to initiation of experimental therapy.

F. Hematological eligibility parameters:

* Granulocyte count greater than or equal to 1,500/mm(3).
* Platelet count greater than or equal to 100,000/mm(3)
* Hgb (Hemoglobin) greater than or equal to 9 Gm/dL
* Lymphocyte count greater than or equal to 500/mm(3).

G. Biochemical eligibility parameters (within 16 days of starting therapy)

-Hepatic function: Bilirubin less than or equal to 1.5 mg/dl, OR patients with Gilbert's syndrome, a total bilirubin less than or equal to 3.0 mg/dL, AST (aspartate aminotransferase) and ALT (alanine aminotransferase) less than 2.5 times upper limit of normal

H. No other active malignancies within the past 3 years (with the exception of non-melanoma skin cancers or carcinoma in situ of the bladder) or life threatening illnesses.

I. Willing to travel to the NIH for follow-up visits.

J. 18 years of age or greater.

K. Able to understand and sign informed consent.

L. Must agree to use effective birth control (such as a condom) or abstinence during and for a period of 4 months after the last vaccination therapy. Patients must be willing to remain on chemical castration therapy, unless they have had surgical castration.

M. Patients must have recovered from acute toxicities related to prior therapy or surgery.

N. Parameters for assessment of baseline renal function:

Serum creatinine less than or equal to 1.5 times the upper limit of normal OR creatinine clearance on a 24-h urine collection of greater than or equal to 60 mL/min.

EXCLUSION CRITERIA:

A. Patients should have no evidence of being immunocompromised as listed below.

* Human immunodeficiency virus positivity due to the potential for decreased tolerance and may be at risk for severe side effects.
* Concurrent use of topical steroids (including steroid eye drops) or systemic steroids. Nasal or inhaled steroid use is permitted.
* Patients who have undergone allogenic peripheral stem cell transplantation or solid organ transplantation requiring immunosuppression.

B. Patients who test positive for active Hepatitis B or Hepatitis C infection.

C. Patients should have no autoimmune diseases that have required treatment such as, Addison's disease, Hashimoto's thyroiditis, or systemic lupus erythematous, Sjogren syndrome, scleroderma, myasthenia gravis, Goodpasture syndrome, active Grave's disease.

D. History of allergy or untoward reaction to prior vaccination with vaccinia virus or to any component of the vaccinia vaccine regimen.

E. Do not administer the recombinant vaccinia vaccine if the recipient, or for at least three weeks after vaccination, their close household contacts (close household contacts are those who share housing or have close physical contact) are: persons with active or a history of eczema or other eczematoid skin disorders; those with other acute, chronic or exfoliative skin conditions (e.g., atopic dermatitis, burns, impetigo, varicella zoster, severe acne, or other open rashes or wounds) until condition resolves; pregnant or nursing women; children 3 years of age and under; and immunodeficient or immunosuppressed persons (by disease or therapy), including HIV (human immunodeficiency virus) infection.

F. Serious intercurrent medical illness (e.g., one that requires treatment) which would interfere with the ability of the patient to carry out the treatment program, including, but not limited to, inflammatory bowel disease, Crohn's disease, ulcerative colitis, or active diverticulitis.

G. Patients with cardiac disease that have fatigue, palpitation, dyspnea or angina with ordinary physical activity (New York Heart Association class 2 or greater) are not eligible.

H. Patients with a history of congestive heart failure or who have objective evidence of congestive heart failure by physical exam or imaging are not eligible.

I. Patients with pulmonary disease that have fatigue or dyspnea with ordinary physical activity are not eligible.

J. Concurrent chemotherapy.

K. No known brain metastasis, or with a history of seizures, encephalitis, or multiple sclerosis.

L. Patients with a serious hypersensitivity reaction to egg products are not eligible.

M. Prior splenectomy.

N. Patients who have received prior flutamide therapy in the last year. (Patients treated with flutamide in the neoadjuvant or adjuvant setting or those previously treated with flutamide who did not have a rising PSA on treatment would be allowed to enroll on the protocol.)

Ages: 18 Years to 110 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2007-02-23 (Actual); Primary Completion 2017-04-27 (Actual); Study Completion 2017-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ravi A Madan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (3):
- United States (3):
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jemal A, Murray T, Ward E, Samuels A, Tiwari RC, Ghafoor A, Feuer EJ, Thun MJ. Cancer statistics, 2005. CA Cancer J Clin. 2005 Jan-Feb;55(1):10-30. doi: 10.3322/canjclin.55.1.10. PMID 15661684
- [Background] Therasse P, Arbuck SG, Eisenhauer EA, Wanders J, Kaplan RS, Rubinstein L, Verweij J, Van Glabbeke M, van Oosterom AT, Christian MC, Gwyther SG. New guidelines to evaluate the response to treatment in solid tumors. European Organization for Research and Treatment of Cancer, National Cancer Institute of the United States, National Cancer Institute of Canada. J Natl Cancer Inst. 2000 Feb 2;92(3):205-16. doi: 10.1093/jnci/92.3.205. PMID 10655437
- [Background] Dillioglugil O, Leibman BD, Kattan MW, Seale-Hawkins C, Wheeler TM, Scardino PT. Hazard rates for progression after radical prostatectomy for clinically localized prostate cancer. Urology. 1997 Jul;50(1):93-9. doi: 10.1016/S0090-4295(97)00106-4. PMID 9218025
- [Derived] Madan RA, Bilusic M, Stein MN, Donahue RN, Arlen PM, Karzai F, Plimack E, Wong YN, Geynisman DM, Zibelman M, Mayer T, Strauss J, Chen G, Rauckhorst M, McMahon S, Couvillon A, Steinberg S, Figg WD, Dahut WL, Schlom J, Gulley JL. Flutamide With or Without PROSTVAC in Non-metastatic Castration Resistant (M0) Prostate Cancer. Oncologist. 2023 Jul 5;28(7):642-e561. doi: 10.1093/oncolo/oyad058. PMID 37134294
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2007-C-0107.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Primary focus of this study compares flutamide with/without vaccine. While patients could get vaccine alone after flutamide progression, this was not a primary focus of the study. With only 11 patients, this group was an exploratory endeavor and there was no statistical plan for comparison to the primary groups.
Groups:
- Flutamide + Vaccine + Sargramostim: Patients receive flutamide orally 3 times a day on days 1-28. Patients also receive recombinant vaccinia PSA vaccine subcutaneously (SC) on day 1 of course 1 only and recombinant fowlpox PSA vaccine SC on day 1 of all subsequent courses. Patients receive sargramostim (GM-CSF) SC on days 1-4. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity. After 3 months of treatment, patients who do not develop clinical progression, but develop biochemical recurrence (e.g., rising PSA levels), discontinue flutamide but may continue to receive vaccine treatment.
  Sargramostim (GM-CSF, Leukine): A recombinant human granulocyte-macrophage colony stimulating factor (GM-CSF) produced by recombinant DNA technology in yeast Saccharomyces cerevisiae). Sargramostim is a 127 amino acid glycoprotein, altered from the native, natural human GM-CSF molecule; the position 23 arginine has been replaced with a leucine to facilitate the expression of the protein in yeast
Period: Initial Drug Administration
Arm/Group | Flutamide Alone | Flutamide + Vaccine + Sargramostim
Started | 33 | 31
Completed | 33 | 31
Not Completed | 0 | 0
Period: Progressed to Receive Vaccine Alone
Arm/Group | Flutamide Alone | Flutamide + Vaccine + Sargramostim
Started | 11 | 0
Completed | 11 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Flutamide Alone | Flutamide + Vaccine + Sargramostim | Total
Number analyzed (Participants) | 33 | 31 | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 7 | 15
  >=65 years | 25 | 24 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.82 (8.61) | 69.84 (8.87) | 70.83 (8.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 33 | 31 | 64
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 31 | 30 | 61
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 5 | 11
  White | 27 | 26 | 53
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 33 | 31 | 64

OUTCOME MEASURES:

1. Primary Outcome: Time to Treatment Failure
Description: Time to treatment failure is defined as a rising Prostatic Specific Antigen (PSA) (Bubley criteria, JCO 1999), development of metastatic disease, or removal from treatment due to excessive toxicity) compared to patients receiving flutamide alone. Normal PSA is 4.0 ng/mL or lower.
Time Frame: Median Potential Follow-up of 46.7 months
Population: Although patients without radiographic progression were allowed to get vaccine after progression on flutamide, the primary comparison in the two groups of this study was Flutamide alone vs. Fluatmiade + vaccine simultaneously. Thus the data on TTF presented is for progression on flutamide alone.
Measure: Median (Full Range); unit: Months
Groups:
- Flutamide + Vaccine + Sargramostim: Patients receive flutamide orally 3 times a day on days 1-28. Patients also receive recombinant vaccinia PSA vaccine subcutaneously (SC) on day 1 of course 1 only and recombinant fowlpox PSA vaccine SC on day 1 of all subsequent courses. Patients receive sargramostim (GM-CSF) SC on days 1-4. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity. After 3 months of treatment, patients who do not develop clinical progression, but develop biochemical recurrence (e.g., rising PSA levels), discontinue flutamide but may continue to receive vaccine treatment.
  Sargramostim (GM-CSF, Leukine): A recombinant human granulocyte-macrophage colony stimulating factor (GM-CSF) produced by recombinant deoxyribonucleic acid (DNA) technology in yeast Saccharomyces cerevisiae).
Arm/Group | Flutamide Alone | Flutamide + Vaccine + Sargramostim
Number analyzed (Participants) | 33 | 31
Months | 4.5 [2 to 70] | 6.9 [2.5 to 40]

2. Secondary Outcome: Count of Participants With Serious and Non-serious Adverse Events Assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0)
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Median Potential Follow-up of 46.7 months
Measure: Count of Participants; unit: Participants
Groups:
- Vaccine Alone After Flutamide: May receive vaccine treatment after flutamide is discontinued.
Arm/Group | Flutamide Alone | Flutamide + Vaccine + Sargramostim | Vaccine Alone After Flutamide
Number analyzed (Participants) | 33 | 31 | 11
Participants | 33 | 31 | 11

3. Secondary Outcome: Number of Participants With Prostatic Specific Antigen (PSA) Response
Description: Complete response is PSA <0.2 confirmed by a second reading at least 4 weeks later. All patients with a PSA decline of >50% (confirmed by a second value at least 4 weeks after the first) and who have no other evidence of disease progression will be reported with both PSA decline only and PSA decline and stable disease on scans. A 25% increase in PSA over nadir is progressive disease with or without evidence of metastatic disease, and/or development of disease on scans or a second occurrence of rising PSA levels in the absence of clinical progression.
Time Frame: Median potential follow-up for all patients is 46.7 months
Population: Although patients without radiographic progression were allowed to get vaccine after progression on flutamide, the primary comparison in the two groups of this study was Flutamide alone vs. Fluatmiade + vaccine simultaneously.
Measure: Count of Participants; unit: Participants
Arm/Group | Flutamide Alone | Flutamide + Vaccine + Sargramostim
Number analyzed (Participants) | 33 | 31
Participants | 7 | 7

4. Secondary Outcome: Percentage of Participants With Antigen Specific Immune Responses Against Prostatic Specific Antigen (PSA)
Description: Antigen specific responses were evaluated using intracellular cytokine staining of cluster of differentiation 4 (CD4) and cluster of differentiation 8 (CD8) cells (evaluating cluster of Differentiation 107a (CD107a), INFg, Interleukin-2 (IL-2), and tumor necrosis factor (TNF) for CD4+ and CD8+ T-cells. Peripheral blood mononuclear cells were separated by Ficoll-Hypaque density gradient separation, washed three times, and preserved in 90% heat-inactivated human A and B blood-type antigens) AB serum and 10% Dimethyl sulfoxide (DMSO) in liquid nitrogen at a concentration of 1 × 10^7 cells/mL until assayed. Analysis of antigen-specific responses following therapy was assessed by intracellular cytokine staining following a period of in vitro stimulation with overlapping 15-mer peptide pools. A more complete description can be found at Heery CR et al, Cancer Immunol Res. 2015 Nov;3(11):1248-56.
Time Frame: 3 months
Measure: Number; unit: percentage of participants
Groups:
- Flutamide + Vaccine + Sargramostim: Patients receive flutamide orally 3 times a day on days 1-28. Patients also receive recombinant vaccinia PSA vaccine subcutaneously (SC) on day 1 of course 1 only and recombinant fowlpox PSA vaccine SC on day 1 of all subsequent courses. Patients receive sargramostim (GM-CSF) SC on days 1-4. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity. After 3 months of treatment, patients who do not develop clinical progression, but develop biochemical recurrence (e.g., rising PSA levels), discontinue flutamide but may continue to receive vaccine treatment.S argramostim (GM-CSF, Leukine): A recombinant human granulocyte-macrophage colony stimulating factor (GM-CSF) produced by recombinant deoxyribonucleic acid (DNA) technology in yeast Saccharomyces cerevisiae). Sargramostim is a 127 amino acid glycoprotein, altered from the native, natural human GM-CSF molecule; the position 23 arginine has been replaced with a leucine to facilitate the expression
Arm/Group | Flutamide Alone | Flutamide + Vaccine + Sargramostim
Number analyzed (Participants) | 19 | 18
percentage of participants | 58 | 56

ADVERSE EVENTS:
Time Frame: Median Potential Follow-up of 46.7 months
Groups:
- Flutamide Alone: Patients receive flutamide orally 3 times a day on days 1-28. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity. After 3 months of treatment, patients who do not develop clinical progression, but develop biochemical recurrence (e.g., rising prostatic specific antigen (PSA) levels) without metastatic disease (as evidenced on scans), as defined in arm II beginning 4 weeks after flutamide therapy is discontinued.
  Flutamide (Eulexin): Orally administered, nonsteroidal, competitive antagonist of testosterone and other androgens at androgenic receptors and may alter the nuclear translocation of the androgen/receptor complex.
Arm/Group | Flutamide Alone | Flutamide + Vaccine + Sargramostim | Vaccine Alone After Flutamide
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/31 | 0/11
Serious Adverse Events (participants affected / at risk) | 4/33 | 5/31 | 0/11
Other Adverse Events (participants affected / at risk) | 32/33 | 29/31 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Flutamide Alone (N=33) | Flutamide + Vaccine + Sargramostim (N=31) | Vaccine Alone After Flutamide (N=11)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Anaphylaxis (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Aortic valve disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac disorders - Other, valvular heart disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 1 (2) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (7) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Mitral valve disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary valve disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Renal and urinary disorders - Other, hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Transient ischemic attacks (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Flutamide Alone (N=33) | Flutamide + Vaccine + Sargramostim (N=31) | Vaccine Alone After Flutamide (N=11)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 10 (17) | 14 (26) | 0 (0)
Alkaline phosphatase increased (Investigations) | 2 (2) | 2 (5) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (3) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 13 (28) | 14 (25) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 3 (4) | 0 (0) | 1 (1)
Aortic valve disease (Cardiac disorders) | 1 (2) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (4) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 9 (11) | 11 (15) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 4 (5) | 1 (1)
Blood bilirubin increased (Investigations) | 3 (3) | 0 (0) | 1 (1)
Blood and lymphatic system disorders - Other, eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Bone infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (2) | 1 (1)
Bronchial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
CD4 lymphocytes decreased (Investigations) | 6 (17) | 3 (7) | 2 (2)
Cardiac disorders - Other, specify (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0) — Lt atrial enlargement; Tachypnea; Coronary disease
Cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 2 (2) | 0 (0)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 5 (6) | 3 (3) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (7) | 5 (6) | 0 (0)
CPK increased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Creatinine increased (Investigations) | 9 (22) | 9 (13) | 2 (2)
Cystitis noninfective (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 7 (12) | 6 (14) | 0 (0)
Dizziness (Nervous system disorders) | 4 (7) | 3 (3) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (6) | 1 (1)
Ear and labyrinth disorders - Other, decreased hearing (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 3 (4) | 3 (4) | 2 (2)
Eye disorders - Other, cataract (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Fever (General disorders) | 0 (0) | 1 (4) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (4) | 0 (0) | 0 (0)
Fatigue (General disorders) | 12 (13) | 16 (31) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0)
Flu like symptoms (General disorders) | 3 (4) | 10 (16) | 3 (4)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 3 (4) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, GI disorder, colon polyps (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gynecomastia (Reproductive system and breast disorders) | 1 (1) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 3 (5) | 2 (3) | 1 (2)
Hematuria (Renal and urinary disorders) | 4 (4) | 6 (9) | 1 (1)
Hemoglobinuria (Renal and urinary disorders) | 4 (4) | 2 (2) | 3 (3)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hot flashes (Vascular disorders) | 5 (5) | 2 (2) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 4 (8) | 4 (7) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 15 (30) | 17 (34) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 6 (11) | 12 (20) | 2 (3)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (3) | 3 (4) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 6 (14) | 7 (9) | 0 (0)
Hypertension (Vascular disorders) | 1 (2) | 0 (0) | 1 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 7 (13) | 6 (9) | 3 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (3) | 3 (4) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 5 (6) | 5 (11) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 2 (3) | 6 (15) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 4 (12) | 5 (13) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 11 (51) | 23 (175) | 11 (51)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Investigations - Other, Bicarbonate, serum-low (Investigations) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 14 (49) | 15 (36) | 5 (10)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Mitral valve disease (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Mucosal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) — Muscle twitching
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 4 (4) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 3 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (6) | 2 (2) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (6) | 1 (1) | 1 (1)
Pain (General disorders) | 4 (6) | 6 (9) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (7) | 5 (6) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 3 (9) | 6 (12) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 8 (18) | 9 (17) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Pulmonary valve disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Renal and urinary disorders - Other, URI (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) — Congestion
Rhinitis infective (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 2 (2) | 2 (5) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0) | 2 (2) — Brittle nails; dermatology/skin- other: cellulitis; dry skin; well differentiated squamous cell carcinoma
Skin induration (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) — Urethral meatus dilatation surgery
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Trismus (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (2) | 3 (5) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 3 (3) | 4 (5) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Urinary retention (Renal and urinary disorders) | 2 (4) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Urine discoloration (Renal and urinary disorders) | 4 (4) | 2 (3) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Weight loss (Investigations) | 1 (1) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 9 (22) | 13 (25) | 2 (6)
Cardiac disorders - Other, specify (Cardiac disorders) | 0 (0) | 2 (3) | 0 (0) — CAD; Tachypnea; Valvular heart disease
Eye disorders - Other, ocular/visual floaters (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Renal and urinary disorders - Other (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (4) | 0 (0) — Erythema left groin; scalp abrasion; lesion, right side of face; right wrist erythema
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 2 (2) | 0 (0) | 0 (0) — Carotid endartectomy cystoscopy, biopsy

LIMITATIONS AND CAVEATS:
Eleven patient cross-over group have no statistical plan in the protocol for analysis, highlighting their exploratory nature.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-04-05): https://cdn.clinicaltrials.gov/large-docs/63/NCT00450463/Prot_SAP_ICF_000.pdf